CLINICAL TRIAL: NCT07038798
Title: Feasibility and Tolerability of Deep Repetitive Transcranial Magnetic Stimulation for Mild Neurocognitive Disorder in Older Adults: A Pilot Study (DeepMIND)
Brief Title: Deep rTMS for Mild Neurocognitive Disorder in Older Adults
Acronym: Deep MIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Dante Duarte, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18440
Record Dates: First submitted 2025-06-02; First posted 2025-06-26 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-05

CONDITIONS: Mild Neurocognitive Disorder
Keywords: Mild Neurocognitive Disorder; Mild NCD; Mild Cognitive Impairment; Deep Transcranial Magnetic Stimulation; deep TMS; dTMS; H coil; H-coil; H1-coil; H4-coil; H7-coil
MeSH Terms: conditions — Neurocognitive Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: One way three-group between-subjects open-label, parallel-arm design
Masking Description: This is an open-label trial. Only study staff processing and analyzing the data will be fully blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active H1-coil dTMS treatment (Experimental): This arm will receive dTMS treatment through active H1-coil.
  Interventions: Device: Brainsway H1-Coil Deep TMS System
- Active H4-coil dTMS treatment (Experimental): This arm will receive dTMS treatment through active H4-coil.
  Interventions: Device: Brainsway H4-Coil Deep TMS System
- Active H7-coil dTMS treatment (Experimental): This arm will receive dTMS treatment through active H7-coil.
  Interventions: Device: Brainsway H7-Coil Deep TMS System

INTERVENTIONS:
Device: Brainsway H1-Coil Deep TMS System — Participants assigned to this arm will complete a 6-week course of 20 dTMS stimulation session using the Brainsway H1-coil.
  Arms: Active H1-coil dTMS treatment
Device: Brainsway H4-Coil Deep TMS System — Participants assigned to this arm will complete a 6-week course of 20 dTMS stimulation session using the Brainsway H4-coil.
  Arms: Active H4-coil dTMS treatment
Device: Brainsway H7-Coil Deep TMS System — Participants assigned to this arm will complete a 6-week course of 20 dTMS stimulation session using the Brainsway H7-coil.
  Arms: Active H7-coil dTMS treatment

SUMMARY:
This study aims to: (1) assess the feasibility and tolerability of three deep transcranial magnetic stimulation (dTMS) coils H1, H4, and H7 in older adults with mild neurocognitive disorder (mild NCD); and (2) evaluate changes in cognition through neuropsychological testing, brain activity through EEG, and mood and sleep through self-report questionnaires. Participants will be assigned to one of three arms: H1- coil vs. H4-coil vs. H7-coil, and all participants will complete assessments examining dTMS side effects, mental health symptoms, and cognition. EEG, questionnaires, and CNS vital signs will be measured at baseline, midpoint (after 10th session- before dTMS treatment on visit 11), and end point, as well as follow up. Collectively, the study will address the absolute and differential feasibility and tolerability of the H1, H4 and H7 coils to provide preliminary data for a future randomized controlled trial comparing this novel intervention to a sham stimulation (placebo) control.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) is a non-invasive therapeutic technique used to stimulate regions of the brain using magnetic pulses. Repeated TMS delivers sequences of pulses for multiple days in a row and is an approved treatment for several psychiatric conditions. Deep TMS (dTMS) is a new technique that uses modified magnetic Hesed coils (H-coils) to stimulate deeper regions of the brain and has been FDA- and Health Canada-approved for major depressive disorder (MDD), obsessive-compulsive disorder, smoking cessation, and anxious-depression in adults. While some research has demonstrated potential benefits of dTMS for cognitive impairment in Alzheimer's disease and other neurodegenerative conditions, its feasibility and tolerability in mild neurocognitive disorder (mild NCD) remain largely unexplored. This innovative pilot study will examine the feasibility and tolerability (side effects, impacts on mental health and cognition), of three dTMS coils (H1, H4 and H7) in older adults with mild NCD. The H1-coil targets bilateral prefrontal cortices, the H4-coil targets the insula and prefrontal cortex, and the H7-coil targets the medial prefrontal cortex and anterior cingulate cortex. These regions are known to be involved in memory, attention, mood regulation, and executive functioning and implicated in mild NCD.

Using an open-label, parallel design, participants aged 60-90 will be assigned to one of three dTMS coils and will complete a six-week course of 20 stimulation sessions (five sessions per week for the first two weeks, three sessions per week for the next two, and two sessions per week for the final two weeks). Each session will include a brief cognitive "priming" task designed to engage brain regions prior to stimulation. In addition to monitoring side effects and retention rates, the study will measure participants' cognitive performance through neuropsychological testing and assess brain function changes through electroencephalogram (EEG) recordings. EEG will be conducted at baseline, midpoint (after 10th session- before dTMS treatment on visit 11), and end point, as well as follow up to capture changes in neural activity and connectivity. This study will lay critical groundwork for a larger, future randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 60 - 90 years old
* Able to provide informed consent to participate in the study
* Subjective concern of mild decline in cognitive function over the past year
* Mild impairment in cognitive performance
* Preserved independence in everyday activities
* Independently mobile (e.g., participants must be able to get in and out of a chair on their own)
* Participants will be required to be on stable dosages of other psychotropic medications for at least 4 weeks prior to screening

Exclusion Criteria:

* Currently receiving treatment or subjective need for treatment for bipolar I or II disorder; psychotic disorder
* Active suicidal behavior
* Severe depression and/or anxiety
* Other neurological or psychiatric disorders accounting for the cognitive deficits
* Impairment in basic and/or instrumental activities of daily living
* Substance use disorder (other than tobacco use disorder) in the past 3 months before entering the study
* Traditional contraindications to rTMS: Intracranial or metal implants in the head or nearby regions, excluding the mouth, that cannot be safely removed; History of epilepsy or seizures; Active unstable medical condition (recent laboratory and neuroimaging alterations, delirium); Pacemaker and/or implantable cardioverter-defibrillators; current use of bupropion, treatment with equivalent benzodiazepine dose to lorazepam >2 mg/day
* People with severe literacy, visual, or hearing issues that affect the ability to engage in the interviews
* People with recurring migraines or headaches (weekly or more)
* Frequent dizziness/vertigo
* Individuals residing beyond the borders of the Greater Hamilton Area and its neighbouring vicinities

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We will implement a sex equity approach by aiming at a 50/50% rate of male and female but allowing an imbalance of maximum 70/30% from either side.
Enrollment: 30 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility criteria 1: Protocol completion | 6 weeks
  Percentage of intervention sessions completed
Feasibility criteria 2: Retention rate | 6 weeks
  Percentage of participants who complete study once enrolled
Feasibility criteria 3: Screening rates and capacity | 6 weeks
  Number of participants (n) screened; n enrolled as a percentage of n screened monthly
Feasibility criteria 4: Recruitment rate and capacity | 6 weeks
  Total number of participants recruited and enrolled per month.
Feasibility criteria 5: Duration of intervention and assessment processes | 6 weeks
  Compared to estimated times, the actual mean times (in min) from start to finish for each dTMS intervention session and mean time (in hours) from start to finish for each visit.
Feasibility criteria 6: Safety of H-coil dTMS treatment | 6 weeks
  Total number of adverse events reported during the treatment sessions assessed by the Side Effects Questionnaire for dTMS (custom-developed for study). At each dTMS stimulation session, participants will complete a questionnaire to evaluate potential adverse effects of dTMS (headache, neck pain, itching and redness at the site of stimulation) according to a 4-point scale.
Tolerability of H-coil dTMS treatment | 6 weeks
  Percentage of participants withdrawn or terminated following enrollment due to adverse events

SECONDARY OUTCOMES:
Changes from baseline on the Everyday Memory Questionnaire (EMQ) | 6 weeks + one-month follow-up
  The Everyday Memory Questionnaire (EMQ) is a 28-item self-report tool, that will be used to assess the frequency and impact of everyday memory problems. It will be measured at baseline (V1), midpoint (after 10th session - before deep TMS treatment on V11) and end point, as well as follow-up.
Changes from baseline in Neurocognitive Performance measured by the CNS Vital Signs Test Battery | 6 weeks + one-month follow-up
  The CNS Vital Signs is the name of a standardized computerized neurocognitive test battery and not a set of physiological vital signs like heart rate or blood pressure. The assessments within CNS Vital Signs are cognitive domains such as memory, executive function, processing speed, etc., not physiological measurements.
  It will be measured at baseline (V1), midpoint (after 10th session - before deep TMS treatment on V11) and end point, as well as follow-up.
Change from baseline on the Hamilton Depression Rating Scale- 24 item (HDRS-24). | 6 weeks + one-month follow-up
  Symptoms of depression will be assessed with the HDRS- 24 item (a 24-item depression checklist) at multiple visits: at baseline (V1), midpoint (after 10th session - before deep TMS treatment on V11) and end point, as well as follow-up.
Change from baseline on the General Anxiety Disorder- 7 item (GAD-7) | 6 weeks + one-month follow-up
  Symptoms of anxiety will be assessed using this 7-item questionnaire at baseline (V1), midpoint (after 10th session - before deep TMS treatment on V11) and end point, as well as follow-up. Scores of 0-4 indicate minimal anxiety; 5-9: mild anxiety; 10-14: moderate anxiety; and 15 or greater: severe anxiety.
Change from baseline on the Pittsburgh Sleeping Quality Index (PSQI) | 6 weeks + one-month follow-up
  Sleep will be monitored and assessed using the Pittsburgh Sleeping Quality Index (PSQI) at baseline (V1), midpoint (after 10th session - before deep TMS treatment on V11) and end point, as well as follow-up.
Change from baseline on the Patient Health Questionnaire (PHQ - Somatic Symptoms) | 6 weeks + one-month follow-up
  Somatic symptoms will be evaluated using the Patient Health Questionnaire (PHQ) somatic inventory at baseline (V1), midpoint (after 10th session - before deep TMS treatment on V11) and end point, as well as follow-up.
Changes from baseline on the Multifactorial Memory Questionnaire (MMQ) | 6 weeks + one-month follow-up
  The Mulitfactorial Memorial Questionnaire (MMQ) is a self-report tool to evaluate three distinct aspects of memory: satisfaction with memory (MMQ-Satisfaction), the frequency of memory lapses (MMQ-Ability), and the use of memory strategies (MMQ-Strategy). It will be measured at baseline (V1), midpoint (after 10th session - before deep TMS treatment on V11) and end point, as well as follow-up.
Changes from baseline in resting-state EEG | 6 weeks + one-month follow-up
  Using electroencephalography (EEG), we will assess alpha, theta and gamma rhythms in fronto-temporo-parietal region, including assessment of connectivity and coherence. We will additionally measure cross-frequency coupling named theta (4-8Hz)-gamma (>25Hz) phase-amplitude coupling (PAC). We will also investigate phase synchronization in upper theta frequency band between prefrontal and temporal areas. Changes in these EEG parameters will be correlated with changes in mood severity and cognitive status, with a focus on working memory improvements. EEG will be performed before dTMS sessions at baseline (V1), midpoint (after 10th session - before deep TMS treatment on V11) and end point, as well as follow-up, by using a wireless dry electrode portable EEG system (CGX Quick 20r). Resting state connectivity, coherence, PAC, and synchronization assessed by EEG will use standardized data processing pipelines in EEG Lab
Changes from baseline in WHO Quality of Life Questionnaire - BREF (WHOQOL-BREF) | 6 weeks + one-month follow-up
  WHOQOL-BREF will measure quality of life in physical, psychological and social domains. This will be measured at baseline (V1), midpoint (after 10th session - before deep TMS treatment on V11) and end point, as well as follow-up.
Changes from baseline Patient Global Impression of Improvement (PGI-I) | 6 weeks + one-month follow-up
  The PGI-I is a single-item global assessment scale used to measure the patient's perceived improvement following an intervention or treatment. This will be measured at midpoint (V11), end of the treatment (V20) and at one-month follow-up.
Changes from baseline on the Monetary Choice Questionnaire (Delay Discounting) | 6 weeks + one-month follow-up
  Delay discounting task which assess propensity to devalue future rewards by asking participants to choose between an immediate small monetary amount and a delayed larger monetary amount. Rewards are hypothetical. This will be measured at baseline (V1), midpoint (after 10th session - before deep TMS treatment on V11) and end point, as well as follow-up
Changes from baseline in blood biomarkers | 6 weeks + one-month follow-up
  Quantity specific biomarkers associated with neurodegeneration {Brain-derived neurotrophic factor (BDNF), Beta-amyloid ratio (Aβ1-42/Aβ1-40 ratio), Phosphorylated Tau 217 (pTAU-217), Neurofilmament light chain (NfL), Cytokines (IGF-1, VEGF, TGF-β1, MCP-1, IL-18)}, will be analyzed using immunoassays, including enzyme-linked immunosorbent assays (ELISA) and single molecular array (SIMOA) technology. These will be measured at baseline (V1) and at one-month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Peter Boris Centre for Addictions Research, St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada